CLINICAL TRIAL: NCT04305262
Title: Continuous Monitoring of Vital Parameters for Early Detection of Clinical Deterioration in Hospitalized Patients - a Part of the Wireless Assessment of Respiratory and Circulatory Distress (WARD) Project
Brief Title: Continuous Monitoring of Vital Parameters for Early Detection of Clinical Deterioration in Hospitalized Patients
Acronym: WARD
Status: Withdrawn | Type: Observational
Why Stopped: due to COVID-19 is was not possible to complete the study
Sponsor: University Hospital Bispebjerg and Frederiksberg (Other)
Collaborators: Technical University of Denmark (Other); Bispebjerg Hospital (Other); Rigshospitalet, Denmark (Other)
Responsible Party: Principal Investigator, Katja Kjær Grønbæk, MD, PhD-student, University Hospital Bispebjerg and Frederiksberg
Other Study IDs: H-19086056
Record Dates: First submitted 2020-03-09; First posted 2020-03-12 (Actual); Last update posted 2022-01-21 (Actual); Status verified 2022-01

CONDITIONS: Continuous Wireless Vital Parameter Monitoring

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Device: Wireless continuous vital parameter monitoring — The patients included in this study will have continuous, wireless monitoring of vital parameters during the first four days of acute admission

SUMMARY:
For patients admitted to the medical ward, it is often difficult to predict if their clinical condition will deteriorate, however subtle changes in vital signs are usually present 8 to 24 hours before a life-threatening event such as respiratory failure leading to ICU admission, or unanticipated cardiac arrest. Such adverse trends in clinical observations can be missed, misinterpreted or not appreciated as urgent. New continuous and wearable 24/7 clinical vital parameter monitoring systems offer a unique possibility to identify clinical deterioration before patients condition progress beyond the point-of-no-return, where adverse events are inevitable. The WARD project aims to determine the correlation between cardiopulmonary micro events and clinical adverse events during the first four days after hospital admission.

ELIGIBILITY:
Inclusion Criteria:

* Adults >18 years
* Acute hospitalization or discharge from Intensive Care Unit (ICU) after an admission of at least 24 hours.
* Early Warning Score (EWS) ≥4 at least once from admission and until inclusion
* One of the following tentative diagnoses as the primary reason for admission: Pneumonia, Dyspnea, Acute myocardial infarction, heartfailure or sepsis
* Inclusion conversation possible within 12 hours of admission or discharge from ICU

Exclusion Criteria:

* Patients that cannot cooperate
* Patients that cannot give informed consent
* Patients with EWS≥4 that is not of presumed physical origin
* Patients with allergies to plaster or silicone
* Patients with pacemaker or ICD
* Patients with treatment limitations (no resuscitation or no admission to ICU)
* Patients with expected discharge within 24 hours
* Patients that have been included in the WARD-COPD study (H-18026653)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Hospitalized patients at general medical wards, that are in high-risk of deterioration
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2020-03-25 (Estimated); Primary Completion 2020-08-01 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Serious desaturation | more than 10 minutes, within the first four days of acute admission
  SpO2 <85% in 10 consecutive minutes

SECONDARY OUTCOMES:
desaturation | more than 60 minutes, within the first four days of acute admission
  SpO2 <92% in 60 consecutive minutes
tachycardia | one minute within the first four days of admission
  Heartrate >130/min
bradycardia | one minute within the first four days of admission
  heartrate >41/min
tachypnea | one minute within the first four days of admission
  Respiration rate >24/min
bradypnea | one minute within the first four days of admission
  Respiration rate <9/min
hypotension | one measurement within the first four days of admission
  Systolic blood pressure <90 mmHg
hypertension | one measurement wihtin the first four days of admission
  systolic blood pressure >219 mmHg

CONTACTS AND LOCATIONS:
Overall Officials: Christian Meyhoff, MD, PhD, Study Chair — Bispebjerg Hospital; Katja Grønbæk, MD, Principal Investigator — Bispebjerg Hospital

IPD SHARING:
Plan to Share IPD: No